CLINICAL TRIAL: NCT06871579
Title: A Pilot Prospective Study of the Esophageal String Test (EST) for the Diagnosis of Helicobacter Pylori
Brief Title: Study of the Esophageal String Test (EST) for the Diagnosis of Helicobacter Pylori
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10002302; 002302-I
Record Dates: First submitted 2025-03-11; First posted 2025-03-12 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01-21

CONDITIONS: Helicobacter Pylori
Keywords: Helicobacter Pylori; Antibiotic resistance; DIAGNOSTIC TEST
MeSH Terms: interventions — Expressed Sequence Tags

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EnteroTracker(R) EST (Experimental): Esophageal string test device consists of a gelatin-coated capsule with a collection string wrapped inside.
  Interventions: Diagnostic Test: EnteroTracker(R) EST

INTERVENTIONS:
Diagnostic Test: EnteroTracker(R) EST — The device consists of a gelatin-coated capsule with a collection string wrapped inside.

SUMMARY:
Background:

Helicobacter pylori is a bacterium that infects the lining of the stomach and intestines. It can cause peptic ulcers, cancers, and infections. Current methods of diagnosing H. pylori infections have limitations. Researchers want to test a new method of testing for H. pylori.

Objective:

To compare the esophageal string test (EST) to standard tests for detecting H. pylori infection.

Eligibility:

People aged 18 years or older with persistent H. pylori infection.

Design:

Participants will have 3 or 4 clinic visits over 2 to 4 months.

Screening visit: Participants will have a physical exam. They will provide a stool sample.

Baseline visit: Participants will have blood tests. Then they will have the EST: One end of a string will be taped to the outside of their cheek; the other end will be packed into a capsule. Participants will swallow the capsule, and the string will unwind down their throat into their stomach. The string will be left in for at least 1 hour. Then researchers will gently pull out the string. The fluids soaked into the string will be studied. Some participants will be prescribed antibiotics.

Follow-up visit 1: Participants whose H. pylori infection was cured by the antibiotics may leave the study. Those who are still infected will have an endoscopy: A flexible tube will be inserted down the throat and into the stomach. It will take tissue samples from the stomach lining. These participants will then receive antibiotics again.

Follow-up visit 2: The physical exam, blood test, and stool sample will be repeated.

...

DETAILED DESCRIPTION:
Study Description:

Adults with active Helicobacter pylori infection will undergo an esophageal string test (EST). The gastric portion of the string will be used for detection of H. pylori by polymerase chain reaction (PCR), as well as assessment of resistance genes to clarithromycin, levofloxacin, and metronidazole. Participants will be treated per current American Gastroenterological Association (AGA) guidelines. A stool antigen test for H. pylori will be performed 4 weeks after completion of therapy to assess cure. Participants who have failed >=2 courses of therapy will undergo endoscopy with resistance testing per AGA recommendations. Patients will be offered antibiotic therapy based on the EST results and will have a repeat H. pylori stool antigen test 4 weeks after completion of therapy.

Primary Objective:

To assess the sensitivity of the gastric portion of the EST in detecting H. pylori infection.

Secondary Objectives:

To assess the ability of the gastric portion of the EST in detecting antimicrobial resistance to clarithromycin, levofloxacin, and metronidazole.

Primary Endpoint:

Proportion of the study population identified positive for H. pylori in EST eluates by PCR.

Secondary Endpoint:

Detection of H. pylori antibiotic resistance genes in EST eluates.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Aged >=18 years
* Diagnosed with H. pylori infection (by endoscopy, stool antigen, or urea breath testing)
* Agreement to adhere to lifestyle considerations throughout study duration
* Ability of participant to provide informed consent

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy or lactation
* Use of antibiotics with activity against H. pylori within 4 weeks of enrollment
* Inability to swallow pills
* Biopsy-proven high grade dysplastic Barrett s esophagus, active peptic ulcer disease, recent (within 4 weeks) upper GI bleed, and/or history of Zollinger Ellison syndrome or gastric bypass surgery

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of the study population identified positive for H. pylori in EST eluates by PCR. | Baseline
  To assess the sensitivity of the gastric portion of the EST in detecting H. pylori infection.

SECONDARY OUTCOMES:
Detection of H. pylori antibiotic resistance genes in EST eluates. | Baseline
  To assess the ability of the gastric portion of the EST in detecting antimicrobial resistance to clarithromycin, levofloxacin, and metronidazole.

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Klion, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li Y, Lv T, He C, Wang H, Cram DS, Zhou L, Zhang J, Jiang W. Evaluation of multiplex ARMS-PCR for detection of Helicobacter pylori mutations conferring resistance to clarithromycin and levofloxacin. Gut Pathog. 2020 Jul 10;12:35. doi: 10.1186/s13099-020-00373-6. eCollection 2020. PMID 32670416
- [Background] Han X, Yu X, Gao X, Wang X, Tay CY, Wei X, Lai B, Marshall BJ, Zhang X, Chua EG. Quantitative PCR of string-test collected gastric material: A feasible approach to detect Helicobacter pylori and its resistance against clarithromycin and levofloxacin for susceptibility-guided therapy. Helicobacter. 2023 Aug;28(4):e12985. doi: 10.1111/hel.12985. Epub 2023 Apr 17. PMID 37066609
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002302-I.html